CLINICAL TRIAL: NCT03808922
Title: A Phase III Randomized Placebo-Controlled Study to Examine the Efficacy and Safety of DAS181 for the Treatment of Lower Respiratory Tract Parainfluenza Infection in Immunocompromised Subjects
Brief Title: Phase III DAS181 Lower Tract PIV Infection in Immunocompromised Subjects (Substudy: DAS181 for COVID-19): RCT Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAS181-3-01; 2018-004318-16 (EudraCT Number)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Lower Respiratory Tract Infection; Parainfluenza; Immunocompromised; COVID-19
Keywords: Parainfluenza; PIV; Immunocompromised; Lower Respiratory Tract Infection; LRTI; COVID19; SARS-CoV-2; Coronavirus; Ansun
MeSH Terms: conditions — Paramyxoviridae Infections; COVID-19; Coronavirus Infections | interventions — oplunofusp

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 and Cohort 2 Treatment (Experimental): DAS181 4.5mg qd x 7 OR 10 days
  Interventions: Drug: DAS181
- Cohort 1 and Cohort 2 Placebo (Placebo Comparator): Placebo qd x 7 OR 10 days
  Interventions: Drug: Placebo
- Cohort 3 (Experimental): DAS181 4.5mg qd x 7 OR 10 days (≥ 40 kg) DAS181 2.5mg qd x 7 OR 10 days (< 40kg)
  Interventions: Drug: DAS181 OL
- Cohort 4 (Experimental): DAS181 4.5mg qd x 7 OR 10 days
  Interventions: Drug: DAS181 OL
- DAS181 COVID-19 Treatment (Experimental): DAS181 4.5mg q12h x 7 OR 10 days
  Interventions: Drug: DAS181 COVID-19
- DAS181 COVID-19 Placebo (Placebo Comparator): Placebo q12h x 7 OR 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAS181 — DAS181 4.5mg nebulized qd x 7 OR 10 days
  Arms: Cohort 1 and Cohort 2 Treatment
Drug: Placebo — Placebo nebulized qd x 7 OR 10 days
  Arms: Cohort 1 and Cohort 2 Placebo; DAS181 COVID-19 Placebo
Drug: DAS181 COVID-19 — DAS181 4.5mg nebulized q12h/day x 7 OR 10 days
  Arms: DAS181 COVID-19 Treatment
Drug: DAS181 OL — DAS181 4.5mg nebulized qd x 7 OR 10 days ≥ 40kg DAS181 2.5mg nebulized qd x 7 OR 10 days < 40kg
  Arms: Cohort 3; Cohort 4

SUMMARY:
This study will seek to enroll immunocompromised patients with Lower Tract parainfluenza infection.

It also contains a sub-study to enroll patients with severe COVID-19.

DETAILED DESCRIPTION:
Eligible subjects (i.e., those meeting the Inclusion / Exclusion criteria) will be enrolled in one of four cohorts based on the following criteria:

Cohort 1:

All eligible subjects in the PoI who are ≥18 year old subjects with a PIV infection and meet all of the following criteria:

1.1 Meet criteria for being severely immunocompromised 1.2 Prior to the onset of PIV infection, had no ongoing need for oxygen therapy due to a chronic respiratory condition (e.g., COPD, sleep apnea) and are assessed as acutely hypoxemic due to their PIV infection 1.3 At the time of randomization are not on mechanical, bi-level or continuous positive airway pressure (Bi-PAP or CPAP) ventilation 1.4 Have no known concurrent respiratory viral coinfection(s)

Cohort 2:

All eligible subjects in the PoI who are ≥18 year old with a PIV infection (including those with PIV and another SAD-RV) who do not meet one or more of the listed criteria for Cohort 1.

Cohort 3:

All eligible subjects in the PoI who are <18 year old subjects with a PIV infection (including those with PIV and another concurrent SAD-RV). There is no lower age limit for this cohort.

Cohort 4:

All eligible subjects in the PoI with a respiratory infection due to any SAD-RV infection except PIV. Eligible subjects with both PIV and an additional concurrent SAD-RV, will be enrolled for either Cohorts 2 or 3 depending on their age. There is no lower age limit for this cohort.

Sub-Study:

Patients with Severe COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. At the time of randomization, requires supplemental oxygen ≥2 LPM due to hypoxemia.
2. Immunocompromised, as defined by one or more of the following:

   * Received an autologous or allogeneic hematopoietic stem cell transplantation (HSCT) at any time in the past
   * Received a solid organ transplant at any time in the past
   * Has been or is currently being treated with chemotherapy for hematologic malignancies (e.g., leukemia, myeloma, lymphoma) and/or solid tumor malignancies (e.g., lung, breast, brain cancer) at any time in the past
   * Has an immunodeficiency due to congenital abnormality (only applicable to subjects age < 18 years old) or pre-term birth (only applicable to subjects age ≤ 2 years old)
3. Has, within 3 days prior to randomization, a confirmed LRTI with a sialic acid dependent respiratory virus
4. If female, subject must meet one of the following conditions:

   * Not be of childbearing potential or
   * Be of childbearing potential and have a negative urine/serum pregnancy test and agrees to practice an acceptable method of contraception
5. Non-vasectomized males are required to practice effective birth control methods
6. Capable of understanding and complying with procedures as outlined in the protocol
7. Provides signed informed consent prior to the initiation of any screening or study-specific procedures

For COVID-19 sub study:

1. Be ≥18 years of age
2. Provide adequate medical history to permit accurate stratification (but health status may be healthy, high-risk conditions, or immunocompromised).
3. Prior to SARS CoV 2 infection, has the ability to carry out self-care activities of daily living (basic ADL)
4. Have lower respiratory tract infection (LRTI) confirmed by CT imaging, with or without contrast, to involve at least 2 lobes of the lung.
5. Has laboratory-confirmation of the presence of SARS CoV 2 in the respiratory tract by at least one of the following samples
6. Satisfy inclusion criteria #1, 4, 5, 6, 7 of the main study

Exclusion Criteria:

1. Subjects may not be on hospice care or, in the opinion of the investigator, have a low chance of survival during the first 10 days of treatment
2. Subjects with Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), or Alkaline Phosphatase (ALP) ≥3x ULN and Total Bilirubin (TBILI) ≥2x ULN Note: Subjects with ALT/AST/ALP ≥ 3x ULN AND TB ≥2x ULN that have been chronically stable (for >1 year on more than one assessments) due to known liver pathology including malignancy (primary or metastasis), chronic medications, transplantation, or chronic infection will not be excluded
3. Female subjects breastfeeding or planning to breastfeed at any time through 30 days after the last dose of study drug
4. Subjects taking any other investigational drug used to treat pulmonary infection.
5. Psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect subject safety and/or compliance
6. Subjects with known hypersensitivity to DAS181 and/or any of its components
7. Subjects with severe sepsis due to either their baseline SAD-RV infection or a concurrent viral, bacterial, or fungal infection and meet at least one of the following criteria:

   * Has evidence of vital organ failure outside of the lung (e.g., liver, kidney)
   * Requires vasopressors to maintain blood pressure

For COVID-19 sub study:

1. Subjects requiring invasive mechanical, Bi-PAP or CPAP ventilation at randomization.
2. Subjects receiving any other investigational or empiric treatment for SARS-2-CoV (either as part of a clinical trial or under emergency approval (approved agents for the management of symptoms, e.g., fever, are permitted).
3. Subjects who are known HIV-positive (and not undetectable at most recent HIV RNA assessment)
4. Subjects who are currently taking immunomodulating biologics (e.g, interferons, interleukin)
5. Subjects with severe sepsis due to either their SARS-CoV-2 infection or a concurrent viral, bacterial, or fungal infection and meeting at least one of the following criteria:

   * Have evidence of vital organ failure outside of the lung (e.g., liver, kidney)
   * Require vasopressors to maintain blood pressure
6. Subjects meeting exclusion criteria #2, 3, 5 and 6 of the main study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects who Return to Room Air (RTRA) (main study) | by Day 28
  Removal of all oxygen support (with stable SpO2)
Percent of subjects with improved COVID-19 Clinical Status Scale (sub-study) | Day 14

SECONDARY OUTCOMES:
All-cause mortality rate (main study) | at Day 28
Percent of subjects who Return to Room Air (RTRA) (main study) | by Day 21
Time (in days) to RTRA (main study) | Days 10, 14, 21, 28
Percent of subjects who achieve clinical stability (main study) | by Day 28
Percent of subjects discharged (without mortality and hospice) (main study) | by Days 14, 21, 28 and 35
Time (in days) to first hospital discharge (without hospice) (main study) | through Day 35
Total number of inpatient days (main study) | up to Day 35
Baseline SAD-RV infection-related mortality rate (main study) | at Day 28
Baseline SAD-RV infection-related mortality rate (main study) | at Day 35
All-cause mortality rate (main study) | at Day 35
Change in pulmonary function (FEV1% predicted) (main study) | Day 1, Day 7, Day 14, Day 28
Time to improved COVID19 clinical status (Sub-study) | Day 5, Day 10, Day 21, Day 28
Time to RTRA | Day 10, Day 14, Day 21, Day 28
Time to Clinical stability | Day 14, Day 21, Day 28
Time to SARS-CoV-2 RNA in the respiratory specimens being undetectable | Day 5, Day 10, Day 14, Day 21, Day 28
Time to Clinical deterioration | Day 5, Day 10, Day 14, Day 21, Day 28
Time to Discharge from hospital (without readmission before Day 28). | Day 14, Day 21, Day 28
Time to Death (all causes) | Day 14, Day 21, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Li, Study Director — Ansun Biopharma, Inc.
Locations (67):
- United States (49):
  - City of Hope cancer Center, Duarte, California
  - UCLA, Los Angeles, California
  - University of California Davis Health System, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center, University of Miami Health System, Miami, Florida
  - Houston Methodist Hospital, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - Louisiana State University, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Universtiy of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University, Durham, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - The Lindner Center- The Christ Hospital, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's, Fort Worth, Texas
  - Texas Health, Fort Worth, Texas
  - Therapeutic Concepts, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson, Houston, Texas
  - VCU Health System, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Froedtert Medical College Pulmonary Clinic, Milwaukee, Wisconsin
- Australia (4):
  - Westmead Hospital, Sydney, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- China (4):
  - Shanghai Pulmonary Hospital, Yangpu, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - Shulan (Hangzhou) Hospital co., LTD, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Rigshospitalet, Copenhagen, Denmark
- Hôpital Henri Mondor, Créteil, Île-de-France Region, France
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Asan Medical Center, Seoul, Gyeonggi-do
  - Samsung Medical Center, Seoul, Gyeonggi-do
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Gyeonggi-do
- Taiwan (2):
  - National Taiwan University Hospital, Zhongzheng, Taipei City
  - National Cheng Kung University Hospital, Tainan